CLINICAL TRIAL: NCT05911126
Title: A Randomized Double Blinded Placebo-controlled Trial to Compare the Effect of Hyoscine-N-butyl Bromide (HBB) or Celecoxib Administered Alone Versus in Combination to Reduce Pain in Patients Undergoing Office Hysteroscopy.
Brief Title: How to Reduce Pain in Patients Undergoing Office Hysteroscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Senderila Abdulkareem, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD-308-2022
Record Dates: First submitted 2023-06-12; First posted 2023-06-20 (Actual); Last update posted 2023-06-20 (Actual); Status verified 2023-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Celecoxib; beta-Globins; Butylscopolammonium Bromide

STUDY DESIGN:
Intervention Model Description: Participants will be allocated in 3 groups, first group receiving 2 medications, second group receiving 1 medication and placebo and a third group receiving 1 medication placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): (60 participants) will receive two oral tablets of HBB (Buscopan 10 mg, Boehringer Ingelheim) and one capsule of Celecoxib 200 mg (Celebrex 200, Pfizer, USA) simultaneously.
  Interventions: Drug: Celecoxib 200 mg, Hyoscine-N-butyl bromide (HBB), placebo tablet
- Group B (Active Comparator): (60 participants) will receive one oral placebo capsule similar in size, structure, and color to celecoxib and two oral tablets of HBB (Buscopan 10 mg, Boehringer Ingelheim)
  Interventions: Drug: Celecoxib 200 mg, Hyoscine-N-butyl bromide (HBB), placebo tablet
- Group C (Active Comparator): (60 participants) will receive two oral placebo tablets similar in size and color to Buscopan tablet and one capsule of Celecoxib 200 mg (Celebrex ® 200, Pfizer, USA).
  Interventions: Drug: Celecoxib 200 mg, Hyoscine-N-butyl bromide (HBB), placebo tablet

INTERVENTIONS:
Drug: Celecoxib 200 mg, Hyoscine-N-butyl bromide (HBB), placebo tablet — Tablet form received prior to the procedure
  Other Names: (Celebrex ® 200, Pfizer, USA), (Buscopan 10 mg, Boehringer Ingelheim)

SUMMARY:
The aim of this study is to compare the effectiveness and the side effects of hyosine-N- butylbromide (HBB) & Celecoxib administered alone versus in combination reducing pain associated with outpatient hysteroscopy in married female patients aged 18-40 attending the outpatient hysteroscopy clinic of Kasr Al Ainy, Cairo University Hospital.

DETAILED DESCRIPTION:
This study will be a prospective single centre study that shall include 180 women aged 18-40 years from the outpatient hysteroscopy clinic, Kasr Al Ainy Cairo University Hospitals. After a self-introduction, each patient will be explained thoroughly about what the study is all about and its objective. All patients will be subjected to history taking (specially to rule out an contraindications of HBB & Celecoxib), pelvic examination and TVUS.

We will make sure that each of the patients voluntarily agrees to participate in this study for this, we will request each patient to sign a written consent form. She will be told that she can withdraw from the study any time.

Patient will be randomized into 3 groups using 1:1:1 allocation ratio. An independent person will generate the allocation sequence using computer- generated random numbers. Allocation will be concealed using sequentially numbered (1-180) opaque sealed envelopes kept with the attending nurse and enclosing a paper denoting group A, B or C. The sealed envelopes will be kept with the attending nurse.

After the patients signs their written consent, the nurse will pick a random number from the available allocation sequence and will open the envelop to detect to which allocated group the patient should be allocated to without showing it to the patient or the observer. The drugs will be stored in the outpatient clinic pharmacy under tags A, B or C and the patient will be given the drug with a glass of water. Neither the patient nor the physician will be aware of the drug used. All patients will receive the enclosed medication 1 hour before procedure.

We will divide the patients into three groups according to the medication will receive.

Group A (60 participants) will receive two oral tablets of HBB (Buscopan 10 mg, Boehringer Ingelheim) and one capsule of Celecoxib 200 mg (Celebrex 200, Pfizer, USA) simultaneously.

Group B (60 participants) will receive one oral placebo capsule similar in size, structure, and color to celecoxib and two oral tablets of HBB (Buscopan 10 mg, Boehringer Ingelheim)

Group C (60 participants) will receive two oral placebo tablets similar in size and color to Buscopan tablet and one capsule of Celecoxib 200 mg (Celebrex ® 200, Pfizer, USA).

The placebo tablets will be manufactured in the faculty of pharmacy - Cairo University.

The procedure will be done in the lithotomy position with a 30°angle 2.9 mm rigid hysteroscopy with 3.8 mm diagnostic sheath [Karl Storz, Germany]. Vaginoscopic approach will be used for insertion of the hysteroscope in all cases (no use of speculum or tenaculum). All the procedures will be done by the same operator using the same equipment. Natural saline will be used as the distension media for all the patients and the pressure of the will be set at 60 mmHg.

The woman's perception of pain will be assessed for each group on three occasions:

* During the procedure (after the hysteroscope will be introduced in the uterine cavity).
* Immediately after the procedure when the hysteroscope will be withdrawn from the uterus.
* 30 minutes after the completion of the procedure.

Pain will be assessed with the use of a 10 visual analogue scale (VAS). VAS of 0 indicates no pain and VAS of 10 indicates the worst possible pain. To assess the pain during the procedure, the attending nurse will reexplain the scale to the patient and will had the her the VAS ruler. The patient will be asked to mark the point she will think will be corresponding to her pain on the ruler at the specific times mentioned above.

Women will also be asked to report any side effect and will be asked about the general acceptability of the procedure whether it was acceptable, difficult, or inacceptable.

The total procedure time will be recorded in seconds and the ease of procedure (easy or difficult) will be recorded by the operator.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for diagnostic hysteroscopy including infertility, bleeding, suspected intrauterine pathologies (eg polypi, septae)
* Reproductive age 20 - 40yrs.
* Postmenstrual days from D-6 to D-11 of the cycle (except in irregular bleeding)

Exclusion Criteria:

* Menopausal and amenorrheic patients
* Contraindication to office hysteroscopy such as:- pelvic inflammatory disease, marked cervical stenosis, pregnancy
* Previous cervical surgery eg; cauterization and conization
* Patients whose vaginoscopic approach will not be enough and where a tenaculum will be used.
* Patients with peptic ulcers or other contraindications to HBB or celecoxib.
* Patients who will have an office operative procedure will be excluded.
* Patients who will refuse or ask to be excluded from the study after enrollment.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2023-06-13 (Estimated); Primary Completion 2023-10-13 (Estimated); Study Completion 2023-12-13 (Estimated)

PRIMARY OUTCOMES:
Pain during whole procedure | 1 hour
  The pain sensation during the procedure. The level of pelvic pain will be rated according to a 10-point visual analogue scale (VAS).

SECONDARY OUTCOMES:
Post procedural pain | 1 hour
  Immediate pain and post 30-mins pain after the completion of the procedure.
  * Side effects such as nausea, vomiting and epigastric pain.
  * Procedure time and ease of entry as reported by the operator.
  * Overall acceptability of the procedure by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Hussein, MD, Study Chair — Cairo University; Nihal M El-Demiry, MD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No